CLINICAL TRIAL: NCT04931927
Title: Impact of Telehealth on Engagement in Psychotherapy and/or Medication Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has been terminated due to a change in study design. The study is no longer a RCT.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Laura Mufson, Professor of Medical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8143
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Psychiatric Diagnosis
Keywords: anxiety; depression; telehealth; behavioral problems
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders; Depression; Problem Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants are randomized to treatment as usual (TAU)
  Interventions: Behavioral: Treatment as usual (TAU)
- MCI-T (Experimental): Participants are randomized to the Making Connections Intervention-Telehealth (MCI-T) plus treatment as usual (TAU)
  Interventions: Behavioral: Making Connections Intervention-Telehealth (MCI-T); Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Making Connections Intervention-Telehealth (MCI-T) — Single session telehealth engagement intervention plus telehealth treatment as usual (TAU) [MCI-T +TAU]
  Arms: MCI-T
Behavioral: Treatment as usual (TAU) — Telehealth treatment as usual without the single session telehealth engagement intervention

SUMMARY:
In the present study, investigators aim to (1) adapt the Making Connections Intervention (MCI) as an intervention to address telehealth engagement and examine whether this targeted intervention can improve youth engagement in telehealth treatment; and (2) assess attitudes towards help-seeking and therapeutic alliance from both the youth and clinician viewpoint to examine the impact of these factors on engagement in telemental health treatment. Forty adolescent participants ages 12-18 will be randomized to either telehealth treatment as usual (TAU) plus the telehealth Making Connections Intervention (MCI-T) engagement session or telehealth TAU alone and followed for 12 weeks from baseline assessment. All clinicians will receive training in the MCI-T intervention and provide either MCI-T + usual care or usual care only depending on the condition to which the adolescents are randomized. All evaluations and therapy sessions will be done over telehealth platform.

DETAILED DESCRIPTION:
Clinicians who participate in the study may be assigned more than one study case, and therefore will complete measures on each study case. All of the clinicians will receive training in the Making Connections Intervention-Telehealth (MCI-T) intervention. The clinicians will deliver the intervention based on the random assignment of the adolescent participants to a treatment arm. When clinicians provide care to adolescents randomized to the MCI-T condition, they will participate in a monthly consultation over telehealth to review cases to promote adherence and fidelity to the treatment.

ELIGIBILITY:
Inclusion Criteria: Youth Sample

1. Youth ages 12-18 years of age receiving an evaluation in the diagnostic evaluation service, the Diagnostic Evaluation and Stabilization Clinic (DESC), or another clinical service in the outpatient Child Behavioral Health Service at NewYork Presbyterian (NYP) - Morgan Stanley Children's Hospital (MSCH)/ NYP-MSCH.
2. English speaking

Exclusion Criteria: Youth Sample

1. Active Suicidal Ideation with current plan and/or intent that requires a higher level of care than outpatient treatment or treatment in DESC
2. Diagnosis of intellectual disability

Inclusion Criteria: Clinician Sample

1. Work as a clinician in any MSCH Outpatient Behavioral Health Service or DESC
2. Clinician consent
3. English or bilingual in English and Spanish

Exclusion Criteria: Clinician Sample

1. None

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Change in the Working Alliance Inventory (WAI-S) | week 1, week 6, week 12 (post intervention)
  The Working Alliance Inventory (WAI-S) reported by both teen and clinician is a self-report measure used to assess three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Items are rated on a 7-point scale ranging from 1 (never) to 7 (always) for the extent to which each of the given statements describes the youth's experience. A total alliance rating is calculated by summing the ratings of all 12 items and ranges from 12-84, with higher scores reflecting a more positive rating of working alliance. The WAI-S will be used to assess changes in working alliance between participants and clinicians through study completion at the 12-week follow-up assessment. The scale will be completed at week 1 about the prior 1 week, at week 6 about the prior 5 weeks, and at week 12 about the prior 6 weeks (post intervention).
Change in Barriers for Adolescent Seeking Health (BASH) | baseline, week 6, week 12 (post intervention)
  The Barriers for Adolescent Seeking Health (BASH) is a 37-item scale that measures adolescents' barriers to seeking help from mental health professionals. Items are rated on a 3-point scale ranging from 1 (not at all) to 3 (a great deal) for the extent to which and individual experiences help-seeking barriers. A total score is calculated by summing the ratings of all 37 items and ranges from 37-111, with higher scores indicating greater barriers to seeking help from a mental health professional. The BASH will be used to assess changes in adolescents' barriers to seeking help from mental health professionals through study completion at the 12-week follow-up assessment. The scale will be completed at baseline about prior lifetime experiences, at week 6 about the prior 6 weeks, and at week 12 about the prior 6 weeks (post intervention).
Change in Attitudes toward Psychological Help-Seeking Scale (ATPHS) | baseline, week 6, week 12
  The Attitudes toward Psychological Help-seeking Scale (ATPHS) is a 5-item scale that assesses stigma in relation to seeking help for psychological problems. Items are rated on a 4-point scale ranging from 0 (strongly disagree) to 3 (strongly agree) for the extent to which an individual . A total score is calculated by summing the ratings of all 5 items and ranges from 0-20, with higher scores indicating more negative attitudes toward seeking psychological help. The ATPHS will be used to assess changes in youth's attitudes toward seeking psychological help through study completion at 12 week follow-up. The scale will be completed at baseline about the participan's lifetime, at week 6 about the prior 6 weeks, and at week 12 about the prior 6 weeks (post intervention).

SECONDARY OUTCOMES:
Change in Progress of Treatment (POT) | week 6, week 12
  The Progress of Treatment Questionnaire (POT) is a 5-item questionnaire that assesses patient progress throughout treatment. Items are rated on a 5-point scale ranging from 1 (not at all) to 5 (very much) for the extent to which the clinician observes patient progress. A total score is calculated by summing the ratings of all 5 items and ranges from 5-25, with higher scores indicating greater patient progress. The POT will be used to assess changes in participants' progress of treatment through the study completion at the 12-week follow-up assessment. The questionnaire will be completed at week 6 about the prior 6 weeks, and at week 12 about the prior 6 weeks.
Change in Client Satisfaction (CSQ-8) | week 6, week 12
  The Client Satisfaction (CSQ-8) is an 8-item self-report questionnaire that measures client satisfaction with psychological services. Items are rated on various different Likert scales as well as through open-ended questions for the extent to which an individual is satisfied with the psychological services they are receiving. A total score is calculated by summing the ratings of all 8 items and accounting for open-ended responses, with higher scores indicating greater client satisfaction. The CSQ-8 will be used to assess changes in participants' satisfaction with the psychological services they are receiving through the study completion at the 12-week follow-up assessment. The questionnaire will be completed at week 6 about the prior 6 weeks, and at week 12 about the prior 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mufson, Ph.D., Principal Investigator — Columbia University/NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No